CLINICAL TRIAL: NCT02492529
Title: Knowing and Remembering: Cognitive and Neural Influences of Familiarity on Recognition Memory in Early Alzheimer's Disease
Acronym: EPMR-MA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014-A01123-44; 35RC14_9777_EPMR-MA (Other: Rennes University Hospital)
Record Dates: First submitted 2014-11-18; First posted 2015-07-08 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer, Recognition Memory, Mild Cognitive Impairment, fMRI
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy volunteers (Other): 60 old healthy volunteers (aged 25-75) will undergo an inclusion visit in order to check inclusion and non inclusion criteria.
  Then will be performed:
  * Neuropsychological tests
  * Experimental procedure
  Interventions: Other: Neuropsychological tests; Other: Experimental procedure
- Patients with early Alzheimer disease (Experimental): 20 patients (aged 60-75) will undergo an inclusion visit in order to check inclusion and non inclusion criteria.
  Then will be performed:
  * Neuropsychological tests
  * Experimental procedure
  * A cranial MRI
  Interventions: Other: Neuropsychological tests; Device: A cranial MRI; Other: Experimental procedure
- Old healthy volunteers (Experimental): 20 healthy volunteers (aged 60-75) will undergo an inclusion visit in order to check inclusion and non inclusion criteria.
  Then will be performed:
  * Neuropsychological tests
  * Experimental procedure
  * A cranial MRI
  Interventions: Other: Neuropsychological tests; Device: A cranial MRI; Other: Experimental procedure

INTERVENTIONS:
Other: Neuropsychological tests — Scales and tests to evaluate:
  * Global cognitive performance
  * Handedness
  * Memory functions performance
  * Gestural praxis functions performance
  * Lexical and semantic functions performance
  * Executive functions performance
  * Memory disorders
  * Way of life
  * Mood
Device: A cranial MRI
  Arms: Old healthy volunteers; Patients with early Alzheimer disease
Other: Experimental procedure

SUMMARY:
Unrandomized, unblinded, monocentric comparative Functional Magnetic Resonance Imaging study.

DETAILED DESCRIPTION:
Prospective functional Magnetic Resonance Imaging study involving a group of participants with Mild Cognitive Impairment due to AD and a control participants group matched for age, education level, verbal Intelligence Quotient as assessed through the French version of the National Adult Reading Test and income group following National Institute of Statistics and Economics Studies classification.

ELIGIBILITY:
Inclusion Criteria:

Volunteers (pilot phase)

* Aged 25 - 75
* French native speakers
* Right-handed
* Education level equal or superior to primary school leaving certificate
* Free from any medical or psychiatric condition that may impact cognition
* Having given written informed consent

Volunteers (experimental phase)

* Aged 60 - 75
* French native speakers
* Right-handed
* Education level equal or superior to primary school leaving certificate
* Free from any medical or psychiatric condition that may impact cognition
* Having given written informed consent

AD-MCI participants

* Aged 60 - 75
* French native speakers
* Right-handed
* Education level equal or superior to primary school leaving certificate
* Fulfilling criteria for " AD-MCI " (Albert et al., 2011)
* Have been seen in a memory medical center or in Memory Resources and Research Medical Center for cognitive symptoms
* Free from any medical or psychiatric condition that may impact cognition
* Able to understand and consent
* Having given written informed consent

Exclusion Criteria:

MRI contraindications (all participants)

* Claustrophobia
* Wearing of any metal implant such as:

  * Heart pacemaker
  * Iron-magnetic surgical clips
  * Any metallic foreign body in the eye or brain

Other criteria (all participants)

* Significant history of neurological or psychiatric disorders
* Ongoing medication that may affect cognitive performances
* Sensory deficit that may interfere with the experimental design (e.g. uncorrected visual impairment)
* Lack of sufficient cooperation during the cognitive tasks
* Persons under major legal protection and/or deprived of liberty

Other criteria (control participants)

- Global cognitive impairment attested by Mattis Dementia Rating Scale or Mini-Mental State Examination, according to available normative data

Other criteria (AD-MCI participants)

* 7 items modified Hachinski ischemic score > 2 (Hachinski et al., 2012)
* Dementia (McKahn, et al., 2011)

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement of recognition memory accuracy measures under the familiarity condition as compared with the novel condition in the AD-MCI group | 3 months
Significant effect of the familiarity vs novelty condition on the pattern of % BOLD signal change in across the brain in the AD-MCI group | 3 months

SECONDARY OUTCOMES:
Significant group effect on the pattern of % BOLD signal change in across the brain | 3 months
Predictive validity of the brain % BOLD signal change pattern for participants clinical status (i.e. controls vs. AD-MCI) | 3 months
Significant interaction between the kind of familiarity condition (i.e. novel, experimental or pre-experimental) and the estimates of recognition memory processes efficiency (i.e. respective contributions of recollection and familiarity, % correct) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Rennes, France

REFERENCES:
- [Result] Jonin PY, Duche Q, Bannier E, Corouge I, Ferre JC, Belliard S, Barillot C, Barbeau EJ. Building memories on prior knowledge: behavioral and fMRI evidence of impairment in early Alzheimer's disease. Neurobiol Aging. 2022 Feb;110:1-12. doi: 10.1016/j.neurobiolaging.2021.10.013. Epub 2021 Oct 29. PMID 34837869